CLINICAL TRIAL: NCT05576480
Title: Efficacy and Safety of Short-course Radiotherapy Sequential Penpulimab in Combination With CAPEOX in the Neoadjuvant Treatment of Microsatellite Stable Locally Advanced Rectal Cancer: a Single-centre, Single-arm, Phase 2 Study
Brief Title: SCRT Sequential Penpulimab in Combination With CAPEOX in the Neoadjuvant Treatment of MSS Locally Advanced Rectal Cancer
Acronym: SPARC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Zhao Ren, Chief Physicion, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPARC
Record Dates: First submitted 2022-10-08; First posted 2022-10-12 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Rectal Cancer; Locally Advanced
Keywords: Immunotherapy; Neoadjuvant Treatment; Locally Advanced Rectal Cancer; Microsatellite stable
MeSH Terms: conditions — Rectal Neoplasms | interventions — penpulimab; spartalizumab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: This is a two staged, single arm phase II trial of short-course radiotherapy sequential Penpulimab in combination with CAPEOX in the neoadjuvant treatment of microsatellite stable locally advanced rectal cancer. Twenty-three patients will be enrolled in the first phase and if the number of pathological complete remission is ≤ 3, the trial will be terminated; if > 3, the trial will proceed to the second phase and continue to enroll up to 48 patients. Taking into account a 15% abscission rate, the total number of patients enrolled will be 55.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCRT sequential Penpulimab in combination with CAPEOX (Experimental): * Short-course radiotherapy (SCRT) + one dose of immunotherapy in week 1：Radiotherapy once daily at 5Gy, D1-D5 (5×5Gy); Penpulimab, 200mg, intravenous for 60±5min, D6 or D7.
  * Rest at week 2, 4 cycles of chemotherapy (CAPEOX) + immunotherapy from week 3 in cycles of 3 weeks: Capecitabine, 1000 mg/m2 orally, administered twice daily, D1-D14 per cycle; Oxaliplatin, 135 mg/m2, intravenous >2h, administered every cycle D1; Penpulimab, 200 mg, administered intravenously for 60 ± 5 min every cycle D1.
  * Clinical re-staging assessment at the end of neoadjuvant therapy allows for a watch-and-wait strategy if cCR is achieved. If any residual lesions remained, radical rectal cancer surgery would be performed at least 2 weeks after the last dose of capecitabine. Whether post-operative adjuvant treatment is performed and the option of post-operative adjuvant treatment is decided by the investigator.
  Interventions: Radiation: Short-course radiotherapy; Drug: Penpulimab; Drug: CAPEOX; Procedure: TME surgery

INTERVENTIONS:
Radiation: Short-course radiotherapy — 5×5Gy in Week 1
Drug: Penpulimab — Apply once in the first week, then every 3 weeks from the third week for four cycles
  Other Names: PD-1 monoclonal antibody
Drug: CAPEOX — Apply every 3 weeks from week 3 for 4 cycles
  Other Names: Capecitabine and oxaliplatin
Procedure: TME surgery — Patient will receive radical rectal cancer surgery

SUMMARY:
The goal of this phase 2 study is to learn about the efficacy and safety of short-course radiotherapy (SCRT) sequential Penpulimab in combination with CAPEOX in the neoadjuvant treatment of microsatellite stable (MSS) locally advanced rectal cancer. The main question it aims to answer is the role of immune checkpoint inhibitors in the neoadjuvant treatment of MSS rectal cancer. Participants will receive neoadjuvant treatment of SCRT sequential Penpulimab in combination with CAPEOX. Participants will undergo a clinical re-staging assessment at the end of neoadjuvant therapy to determine whether to adopt a watch-and-wait strategy or undergo radical surgery.

DETAILED DESCRIPTION:
Today there has been an outbreak progress in immunotherapy for tumors, where immune checkpoint inhibitors targeting PD-1/PD-L1 have been approved for the treatment of a variety of tumors, bringing long-term benefits to some patients, especially colorectal cancer and other solid tumors with dMMR/MSI-H have been identified as the best indication population for immunotherapy. However, the majority of patients presented with microsatellite stable (MSS) or pMMR status had a low response rate to immunotherapy. How to improve the response to immunotherapy in these patients has been a challenge in the field of colorectal cancer immunotherapy. A number of preclinical and small clinical studies have identified immunotherapy in combination with other treatments such as chemotherapy, radiotherapy, anti-angiogenic drugs and targeted therapies as potentially viable options to overcome immune resistance and improve the outcome of MSS colorectal cancer. Preclinical and small clinical studies have demonstrated that radiotherapy may induce antigen release from tumors with low neoantigen load and activate dendritic cells, thereby activating CD8+ T lymphocyte-mediated anti-cancer immune responses. In patients with locally advanced rectal cancer, neoadjuvant chemoradiotherapy can increase PD-L1 expression in tumor cells, suggesting that the combination of radiotherapy and PD-1/PD-L1 inhibitors may have a synergistic effect. To further improve the treatment outcomes of locally advanced rectal cancer, we designed an exploratory observational study to observe the efficacy and safety of a regimen of short-course radiotherapy combined with chemotherapy and the addition of the PD-1 monoclonal antibody in locally advanced rectal cancer, and to initially explore the feasibility a watch-and-wait strategy for patients with rectal cancer who have reached pCR.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* 18 years < age ≤ 75 years
* ECOG score is 0-1
* Patients with pathologically confirmed rectal adenocarcinoma, assessed by MRI as mid-low rectal cancer (the lower border of the tumor is less than 10cm from the anal verge), clinical stage II-III (cT1-2N1-2M0 or T3-4N0-2M0) according to the 8th Edition of AJCC Cancer Staging Manual
* Without emergency operation due to complication (bleeding, perforation or obstruction) caused by rectal cancer
* Microsatellite Instability detection using PCR capillary electrophoresis results in MSS
* Without any anti-tumor treatment
* No distant metastasis
* Have an imaging measurable or clinically assessable lesion
* Adequate organ and bone marrow function
* Female participants of childbearing age or male participants whose sexual partners are women of childbearing age are required to use effective contraception for the entire treatment period and for 6 months after the end of the treatment period

Exclusion Criteria:

* Recurrent rectal cancer
* Previous treatment with pelvic radiotherapy, rectal cancer surgery, chemotherapy, targeted therapy, immune checkpoint inhibitors (including but not limited to PD-1, PD-L1, CTLA-4)
* Proven inability to receive radiotherapy or allergy to the components of Penpulimab, capecitabine, oxaliplatin or their excipients
* Intestinal obstruction due to tumor (except in patients who have received a stoma)
* History of other primary malignancies, except for: malignancies in complete remission for at least 2 years prior to enrolment and not requiring other treatment during the study period; adequately treated non-melanoma skin cancer or lentigo maligna with no evidence of disease recurrence; adequately treated carcinoma in situ with no evidence of disease recurrence
* Active, known or suspected autoimmune disease or history of this disease within the previous 2 years (patients with vitiligo, psoriasis, alopecia or Graves' disease not requiring systemic treatment within the last 2 years, hypothyroidism requiring only thyroid hormone replacement therapy and type I diabetes requiring only insulin replacement therapy may be enrolled)
* Any of the following within 6 months prior to the start of treatment: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (New York Heart Association classification II-IV), cerebrovascular event, transient ischaemic attack, severe arrhythmia requiring drug treatment or symptomatic pulmonary embolism
* History of allogeneic organ transplantation and allogeneic haematopoietic stem cell transplantation
* Uncontrolled comorbidities including but not limited to: HIV infected; Serious infections that are active or poorly controlled clinically
* Pregnant woman or lactating woman
* Patients who have participated in another drug clinical trial within 4 weeks
* Suffering from acute or chronic active hepatitis B (HBsAg-positive and HBV DNA ≥ 200 IU/mL or ≥ 103 copies/mL) or acute or chronic active hepatitis C (HCV-positive and HCV RNA-positive)
* Received live attenuated vaccine within 4 weeks prior to enrolment or planned during the study period
* Major surgical procedure within 4 weeks prior to enrolment
* History of interstitial pneumonia
* Other acute or chronic diseases, mental disorders, or laboratory test abnormalities that may result in: increasing the risk associated with research participation or drug administration, or interfering with the interpretation of the results of the study, and the patient was classified as not eligible to participate in this study according to the judgment of the researchers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete remission rate (pCR) | One month after surgery
  The proportion of complete remissions detected by postoperative pathological examination (%)

SECONDARY OUTCOMES:
Clinical complete remission rate (cCR) | Three weeks after neoadjuvant therapy
  The proportion of complete remissions detected by imaging, endoscopy and digital rectal examination (%)
Objective response rate (ORR) | One month after surgery
  Sum of proportion in complete and partial remission (%)
3-year disease free survival rate (3y-DFS) | 36 months after surgery
  3-year disease free survival rate estimated based on Kaplan-Meier method
R0 resection rate | One month after surgery
  Histologically complete resection rate (%)
Sphincter preservation rate | One month after surgery
  The proportion of low rectal cancer patients retaining the sphincter in radical surgery (%)
Early morbidity rate | 30 days after surgery
  Morbidity rate 30 days after surgery (%)
Number and severity of adverse events | 36 months after surgery
  Number and severity of adverse events using CTCAE V5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ren Zhao, MD, PHD, Principal Investigator — Ruijin Hospitlal , Shanghai Jiaotong University School of Medicine
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, None Selected, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bahadoer RR, Dijkstra EA, van Etten B, Marijnen CAM, Putter H, Kranenbarg EM, Roodvoets AGH, Nagtegaal ID, Beets-Tan RGH, Blomqvist LK, Fokstuen T, Ten Tije AJ, Capdevila J, Hendriks MP, Edhemovic I, Cervantes A, Nilsson PJ, Glimelius B, van de Velde CJH, Hospers GAP; RAPIDO collaborative investigators. Short-course radiotherapy followed by chemotherapy before total mesorectal excision (TME) versus preoperative chemoradiotherapy, TME, and optional adjuvant chemotherapy in locally advanced rectal cancer (RAPIDO): a randomised, open-label, phase 3 trial. Lancet Oncol. 2021 Jan;22(1):29-42. doi: 10.1016/S1470-2045(20)30555-6. Epub 2020 Dec 7. PMID 33301740
- [Background] Dossa F, Chesney TR, Acuna SA, Baxter NN. A watch-and-wait approach for locally advanced rectal cancer after a clinical complete response following neoadjuvant chemoradiation: a systematic review and meta-analysis. Lancet Gastroenterol Hepatol. 2017 Jul;2(7):501-513. doi: 10.1016/S2468-1253(17)30074-2. Epub 2017 May 4. PMID 28479372